CLINICAL TRIAL: NCT07231029
Title: An Open-label Pharmacokinetic Study of TS-172 in Patients With Hepatic Impairment
Brief Title: A Pharmacokinetic Study of TS-172 in Patients With Hepatic Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS172-03-10
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Patients With Mild or Moderate Hepatic Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Experimental)
  Interventions: Drug: TS-172
- Moderate hepatic impairment (Experimental)
  Interventions: Drug: TS-172
- Normal hepatic function (Experimental)
  Interventions: Drug: TS-172

INTERVENTIONS:
Drug: TS-172 — Single oral administration of TS-172 20mg

SUMMARY:
An open-label study to evaluate the effect of TS-172 administration on pharmacokinetics in patients with hepatic impairment

ELIGIBILITY:
<Inclusion criteria for patients with hepatic impairment>

1. Japanese male and female patients whose age is >=18 and <=75 years at the time of obtaining informed consent
2. Patients with chronic hepatic impairment
3. Patients who were classified by the principal investigator or sub-investigator as Class A (mild) or Class B (moderate) by Child-Pugh classification at the screening test Other protocol defined inclusion criteria could apply.

<Inclusion criteria for subjects with normal hepatic function>

1. Japanese male and female patients whose age is >=18 and <=75 years at the time of obtaining informed consent
2. Subjects whose body mass index is >=18.5 and <35.0 at the screening test Other protocol defined inclusion criteria could apply.

<Exclusion criteria for patients with hepatic impairment>

1. Patients with medical history of liver resection or liver transplantation
2. Patients with grade II or higher hepatic encephalopathy
3. Patients whose eGFR is <45 mL/min/1.73 m2 at screening test Other protocol defined exclusion criteria could apply.

<Exclusion criteria for subjects with normal hepatic function>

1. Subjects with current condition or medical history of diseases that are ineligible for participation in the study
2. Subjects whose eGFR is <60 mL/min/1.73 m2 at screening test Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of unchanged form and metabolites | Up to 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No